CLINICAL TRIAL: NCT07116603
Title: Prevalence of Urinary Incontinence and Identification of Risk Factors Among Female Medical Students
Acronym: UI medical stu
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ismail Biyik, Associate Professor, Kutahya Health Sciences University
Other Study IDs: Kutahya Health Sciences Uni.; Kutahya Health Sciences Uni. (Registry Identifier: Kutahya Health Sciences Uni.)
Record Dates: First submitted 2025-08-06; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Urinary Incontinence
Keywords: Urinary incontinence; medical student
MeSH Terms: conditions — Urinary Incontinence | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical student cohort: Female Medical student in Kütahya Health Sciences University
  Interventions: Diagnostic Test: Questionnaire and Physical Exam

INTERVENTIONS:
Diagnostic Test: Questionnaire and Physical Exam — Participants completed the International Continence Questionnaire-Short Form (ICIQ-SF) and the Incontinence Impact Questionnaire (IIQ-7) form were completed

SUMMARY:
The prevalence of urinary incontinence and risk factors were investigated among female students studying at Kütahya Health Sciences University Faculty of Medicine.

DETAILED DESCRIPTION:
Students who voluntarily participated in the study, had access to the online structured questionnaire distributed via a computer-based system, completed the survey in full, and were actively enrolled during the study period were included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Female Medical Student Speak Turkish

Exclusion Criteria:

* Psychological disorder that impairs understanding

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female
Study Population: Female Medical Student in Kütahya Health Sciences University
Sampling Method: Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Prevelance of urinary incontinence | 1 march 2025 - 1 may 2025
  Prevelance of urinary incontinence was calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya Medical Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The researchers have not yet decided whether to share the study protocol publicly.

REFERENCES:
- [Background] Patel UJ, Godecker AL, Giles DL, Brown HW. Updated Prevalence of Urinary Incontinence in Women: 2015-2018 National Population-Based Survey Data. Female Pelvic Med Reconstr Surg. 2022 Apr 1;28(4):181-187. doi: 10.1097/SPV.0000000000001127. Epub 2022 Jan 12. PMID 35030139